CLINICAL TRIAL: NCT06240741
Title: A Prospective, Open-label, Multi-center, Single Arm, Phase III Study of [68Ga]Ga-DOTA-TATE in the Diagnosis of Patients With Neuroendocrine Neoplasms (NENs) and Healthy Volunteers in Japan
Brief Title: A Prospective, Open-label Study of [68Ga]Ga-DOTA-TATE in Patients With Neuroendocrine Neoplasms (NENs) and Healthy Volunteers in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Eckert & Ziegler Radiopharma GmbH (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAA501A11301
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Neoplasms
Keywords: [68Ga]Ga-DOTA-TATE; Neuroendocrine Neoplasms (NENs); Positron Emission Tomography (PET); Computerized Tomography (CT); PET/CT; Diagnostic performance; Sensitivity; Specificity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-DOTA-TATE (Experimental): All eligible participants will receive [68Ga]Ga-DOTA-TATE via intravenous injection at a dose of 2 MBq/kg (0.054 mCi/kg) of body weight up to a maximum total dose of 200 MBq (5.4 mCi)
  Interventions: Drug: [68Ga]Ga-DOTA-TATE; Drug: 68Ge/68Ga Generator

INTERVENTIONS:
Drug: [68Ga]Ga-DOTA-TATE — Single intravenous injection of [68Ga]Ga-DOTA-TATE determined by body weight (2 Mega-Becquerel (MBq) / kilogram (kg) (0.054 Millicurie (mCi)/kilogram (kg)) of body weight up to a maximum total dose of 200 MBq (5.4 mCi)) at the imaging day (Day 1).
  Other Names: AAA501
Drug: 68Ge/68Ga Generator — Radionuclide generator
  Other Names: EZR001

SUMMARY:
The purpose of this study was to evaluate the diagnostic performance of [68Ga]Ga-DOTA-TATE Positron Emission Tomography (PET)/Computerized Tomography (CT) imaging compared with conventional imaging (CIM) as standard of truth in patients with neuroendocrine neoplasms (NENs) and healthy volunteers (HVs).

The data from this study was collected in order to provide the evidence for diagnosis of [68Ga]Ga-DOTA-TATE PET/CT imaging in patient with NENs in Japan.

DETAILED DESCRIPTION:
A total of 71 participants (48 patients with confirmed/suspected NENs and 23 HVs) were enrolled to ensure that at least 70 participants (47 patients with confirmed/suspected NENs and 23 HVs) were evaluable for the co-primary endpoints. All enrolled participants were administered [68Ga]Ga-DOTA-TATE and PET/CT scan.

The co-primary endpoints of the subject-level sensitivity and the subject-level specificity were assessed by comparing the central reading results of the [68Ga]Ga-DOTA-TATE PET/CT scan to the central reading results of Conventional imaging (CIM).

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent must have been obtained prior to participation in the study
2. Participants must have been adults >= 18 years of age
3. ECOG performance status 0-2
4. For patient with NENs only: Participants were to be confirmed NENs based on histopathology, imaging and other relevant examination, or with suspected NENs which localization could not have been confirmed by CIM
5. For HVs only: Male or female participant in good health condition as determined by no clinically significant findings from medical history, physical examination, vital signs, lab test and ECG
6. Women of childbearing potential must havehad a negative urine or blood pregnancy test.

Key Exclusion Criteria:

1. Inability to complete the needed investigational and conventional imaging due to any reason (severe claustrophobia, inability to lie still for the entire imaging time, etc.)
2. Any additional medical condition, serious intercurrent illness, concomitant cancer or other extenuating circumstance that, in the opinion of the Investigator, would indicate a significant risk to safety or impair study participation
3. Known allergy, hypersensitivity, or intolerance to [68Ga]Ga-DOTA-TATE and [111In]In-Pentetreotide
4. Therapeutic use of any somatostatin analogue except for the following washout period

   * Short-acting analogs of somatostatin can be used up to 24 hours before injection of [68Ga]Ga-DOTA-TATE.
   * Long-acting analogs of somatostatin can be used up to 28 days before injection of [68Ga]Ga-DOTA-TATE.
5. Prior administration of a radiopharmaceutical unless 10 or more half-lives have elapsed before injection of [68Ga]Ga-DOTA-TATE
6. Use of other investigational drugs within 30 days before screening
7. Participants who were pregnant.
8. Participants who were lactating.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Japan (7):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was not designed to compare efficacy between NEN patients and HVs, but rather to assess sensitivity and specificity of Ga-DOTA-TATE PET/CT imaging against the CIM in the population which includes both of CIM positive and negative.
Pre-assignment Details: Therefore, efficacy results related to the diagnostic performance are presented as a single combined population of NEN patients and HVs. Baseline characteristics, other efficacy (e.g. number of lesions), safety, and PK results are presented separately due to the differences between the NEN patient and HV populations.
  These approaches are as per the protocol and the statistical analysis plan.
Groups:
- [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs; Healthy Volunteers: All eligible participants received [68Ga]Ga-DOTA-TATE via intravenous injection at a dose of 2 MBq/kg (0.054 mCi/kg) of body weight up to a maximum total dose of 200 MBq (5.4 mCi)
Period: Overall Study
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Started | 48 | 23
Completed | 48 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers | Total
Number analyzed (Participants) | 48 | 23 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 22 | 51
  >=65 years | 19 | 1 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 25 | 13 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 48 | 23 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of [68Ga]Ga-DOTA-TATE Positive Participants (TP Participants) Among CIM Positive Participants (TP or FN Participants)
Description: Subject-level sensitivity is defined as the proportion of [68Ga]Ga-DOTA-TATE PET/CT imaging positive participants (i.e. TP participants) among CIM positive participants (i.e. TP or FN participants).
  * TP participants were those who showed at least one lesion based on both [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM by central read.
  * FN participants were those who did not show any lesions based on [68Ga]Ga-DOTA-TATE PET/CT imaging but showed at least one lesion based on CIM by central read.
  True Positive [TP] False Positive [FP] False Negative [FN] True Negative [TN]
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact, and who are CIM positive participants (TP or FN participants).
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Confirmed/suspected NENs + HVs. All eligible participants received [68Ga]Ga-DOTA-TATE via intravenous injection at a dose of 2 MBq/kg (0.054 mCi/kg) of body weight up to a maximum total dose of 200 MBq (5.4 mCi)
Arm/Group | All Participants
Number analyzed (Participants) | 46
Participants
  True Positive [TP] | 40
  False Negative [FN] | 6

2. Primary Outcome: Number of [68Ga]Ga-DOTA-TATE Negative Participants (TN Participants) Among CIM Negative Participants (TN or FP Participants)
Description: Subject-level specificity is defined as the proportion of [68Ga]Ga-DOTA-TATE PET/CT imaging negative participants (i.e. TN participants) among CIM negative participants (i.e. TN or FP participants).
  * TN participants were those who did not show any lesions based on both [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM by central read.
  * FP participants were those who showed at least one lesion based on [68Ga]Ga-DOTA-TATE PET/CT imaging but did not show any lesions based on CIM by central read.
  True Positive [TP] False Positive [FP] False Negative [FN] True Negative [TN]
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact, and who are CIM negative participants (TN or FP participants).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 25
Participants
  True Negative [TN] | 23
  False Positive [FP] | 2

3. Primary Outcome: Subject-level Sensitivity
Description: Subject-level sensitivity is defined as the proportion of [68Ga]Ga-DOTA-TATE PET/CT imaging positive participants (i.e. TP participants) among CIM positive participants (i.e. TP or FN participants).
  True Positive [TP] False Positive [FP] False Negative [FN] True Negative [TN]
  Sensitivity = TP / (TP + FN)
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Sensitivity (%)
Arm/Group | All Participants
Number analyzed (Participants) | 46
Sensitivity (%) | 87.0 [73.74 to 95.06]

4. Primary Outcome: Subject-level Specificity
Description: Subject-level specificity is defined as the proportion of [68Ga]Ga-DOTA-TATE PET/CT imaging negative participants (i.e. TN participants) among CIM negative participants (i.e. TN or FP participants).
  True Positive [TP] False Positive [FP] False Negative [FN] True Negative [TN]
  Specificity = TN / (TN + FP).
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Specificity (%)
Arm/Group | All Participants
Number analyzed (Participants) | 25
Specificity (%) | 92.0 [73.97 to 99.02]

5. Secondary Outcome: Number of Participants Who Are Positive on Both [68Ga]Ga-DOTA-TATE PET/CT Imagings and CIM (TP Participants) Among Participants Who Are Positive on [68Ga]Ga-DOTA TATE PET/CT Imaging (TP or FP Participants)
Description: Subject-level positive predictive values (PPV) is defined as the proportion of TP participants among [68Ga]Ga-DOTA-TATE PET/CT imaging positive participants (i.e. TP or FP participants).
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact, and who are positive on [68Ga]Ga-DOTA TATE PET/CT imaging (TP or FP participants).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 42
Participants
  True Positive [TP] | 40
  False Positive [FP] | 2

6. Secondary Outcome: Number of Participants Who Are Negative on Both [68Ga]Ga-DOTA-TATE PET/CT Imaging and CIM (TN Participants) Among Participants Who Are Negative on [68Ga]Ga-DOTA-TATE PET/CT Imaging (TN or FN Participants)
Description: Subject-level NPV was defined as the proportion of TN participants among [68Ga]Ga-DOTA-TATE PET/CT imaging negative participants (i.e. TN or FN participants).
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact, and who are negative on [68Ga]Ga-DOTA-TATE PET/CT imaging (TN or FN participants).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
Participants
  False Negative [FN] | 6
  True Negative [TN] | 23

7. Secondary Outcome: Subject-level PPV
Description: Subject-level positive predictive values (PPV) is defined as the proportion of TP participants among [68Ga]Ga-DOTA-TATE PET/CT imaging positive participants (i.e. TP or FP participants).
  PPV (Subject-level positive predictive values) = TP / (TP + FP)
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact, and who are [68Ga]Ga-DOTA-TATE PET/CT imaging positive participants (i.e. TP or FP participants).
Measure: Number (95% Confidence Interval); unit: PPV (%)
Arm/Group | All Participants
Number analyzed (Participants) | 42
PPV (%) | 95.2 [83.84 to 99.42]

8. Secondary Outcome: Subject-level NPV
Description: Subject-level NPV was defined as the proportion of TN participants among [68Ga]Ga-DOTA-TATE PET/CT imaging negative participants (i.e. TN or FN participants).
  NPV (Subject-level negative predictive values) = TN / (TN + FN)
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact, and who are [68Ga]Ga-DOTA-TATE PET/CT imaging negative participants (i.e. TN or FN participants).
Measure: Number (95% Confidence Interval); unit: NPV (%)
Arm/Group | All Participants
Number analyzed (Participants) | 29
NPV (%) | 79.3 [60.28 to 92.01]

9. Secondary Outcome: Participants Who Have Consistent Results (i.e. TP or TN Participants) Among All Participants Assessed by [68Ga]Ga-DOTA-TATE PET/CT Imaging and CIM - Subject-level Accuracy
Description: Subject-level accuracy is defined as the proportion of TP and TN participants among all patients in the EFF (i.e. TP+TN+FP+FN participants).
  Accuracy = (TP + TN) / (TP + TN + FP + FN).
Time Frame: Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM. HVs had to have results of [68Ga]Ga-DOTA-TATE PET/CT imaging, with a valid measurement without a protocol deviation with impact.
Measure: Number (95% Confidence Interval); unit: Accuracy (%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
Accuracy (%) | 88.7 [79.00 to 95.01]

10. Secondary Outcome: Region-level Sensitivity
Description: Region-level sensitivity is defined as the proportion of [68Ga]Ga-DOTA-TATE PET/CT imaging positive regions (TP regions) among CIM positive regions (i.e. TP or FN regions).
  Sensitivity = TP / (TP + FN)
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Sensitivity (%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
Sensitivity (%)
  Liver: number analyzed (Participants) | 36
  Liver | 77.8 [60.85 to 89.88]
  Pancreas: number analyzed (Participants) | 14
  Pancreas | 42.9 [17.66 to 71.14]
  Gastrointestinal tract: number analyzed (Participants) | 1
  Gastrointestinal tract | 0 [0 to 97.50]
  Lymph nodes: number analyzed (Participants) | 16
  Lymph nodes | 75.0 [47.62 to 92.73]
  Other: number analyzed (Participants) | 13
  Other | 84.6 [54.55 to 98.08]

11. Secondary Outcome: Region-level Specificity
Description: Region-level specificity is defined as the proportion of [68Ga]Ga-DOTA-TATE PET/CT imaging negative regions (TN regions) among CIM negative regions (i.e. TN or FP regions).
  Specificity = TN / (TN + FP)
  Note: Even when a participant is categorized as positive in subject-level, he/she can still have negative results in region-level. e.g. When only Liver is positive and other regions are negative, the participant is categorized as positive in subject-level. As all participants had at least one CIM-negative region and were included in the table, the number of participants analyzed is 71.
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Specificity(%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
Specificity(%)
  Liver: number analyzed (Participants) | 35
  Liver | 97.1 [85.08 to 99.93]
  Pancreas: number analyzed (Participants) | 57
  Pancreas | 89.5 [78.48 to 96.04]
  Gastrointestinal tract: number analyzed (Participants) | 70
  Gastrointestinal tract | 95.7 [87.98 to 99.11]
  Lymph nodes: number analyzed (Participants) | 55
  Lymph nodes | 83.6 [71.20 to 92.23]
  Other: number analyzed (Participants) | 58
  Other | 94.8 [85.62 to 98.92]

12. Secondary Outcome: Region-level Positive Predictive Values (PPV)
Description: Region-level PPV is defined as the proportion of regions which are positive on both [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM (TP regions) among [68Ga]Ga-DOTA-TATE PET/CT imaging positive regions (i.e. TP or FP regions).
  Region-level positive predictive values (PPV) = TP / (TP +FP)
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: PPV (%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
PPV (%)
  Liver: number analyzed (Participants) | 29
  Liver | 96.6 [82.24 to 99.91]
  Pancreas: number analyzed (Participants) | 12
  Pancreas | 50.0 [21.09 to 78.91]
  Gastrointestinal tract: number analyzed (Participants) | 3
  Gastrointestinal tract | 0 [0 to 70.76]
  Lymph nodes: number analyzed (Participants) | 21
  Lymph nodes | 57.1 [34.02 to 78.18]
  Other: number analyzed (Participants) | 14
  Other | 78.6 [49.20 to 95.34]

13. Secondary Outcome: Region-level Negative Predictive Values (NPV)
Description: Region-level NPV is defined as the proportion of regions which are negative on both [68Ga]Ga- DOTA-TATE PET/CT imaging and CIM (TN regions) among [68Ga]Ga-DOTA-TATE PET/CT imaging negative regions (i.e. TN or FN regions).
  Region-level negative predictive values (NPV) = TN / (TN + FN)
  Note: Even when a participant is categorized as positive in subject-level, he/she can still have negative results in region-level. e.g. When only Liver is positive and other regions are negative, the participants is categorized as positive in subject-level. As all participants had at least one negative region by Ga-DOTA-TATE PET/CT and were included in the table, the number of participants analyzed = 71.
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: NPV (%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
NPV (%)
  Liver: number analyzed (Participants) | 42
  Liver | 81.0 [65.88 to 91.40]
  Pancreas: number analyzed (Participants) | 59
  Pancreas | 86.4 [75.02 to 93.96]
  Gastrointestinal tract: number analyzed (Participants) | 68
  Gastrointestinal tract | 98.5 [92.08 to 99.96]
  Lymph nodes: number analyzed (Participants) | 50
  Lymph nodes | 92.0 [80.77 to 97.78]
  Other: number analyzed (Participants) | 57
  Other | 96.5 [87.89 to 99.57]

14. Secondary Outcome: Region-level Accuracy
Description: Region-level accuracy is defined as the proportion of regions which are CIM and [68Ga]Ga-DOTA-TATE PET/CT imaging positive (TP regions) or negative (TN regions) among regions detected by CIM and [68Ga]Ga-DOTA-TATE PET/CT imaging (i.e. TP+TN+FP+FN regions).
  Accuracy = (TP + TN) / (TP + TN + FP + FN).
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: accuracy (%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
accuracy (%)
  Liver | 87.3 [77.30 to 94.04]
  Pancreas | 80.3 [69.14 to 88.78]
  Gastrointestinal tract | 94.4 [86.20 to 98.44]
  Lymph nodes | 81.7 [70.73 to 89.87]
  Other | 93.0 [84.33 to 97.67]

15. Secondary Outcome: Region-level True Positive
Description: TP regions were the regions which showed at least one lesion based on both [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM by central read
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Participants
  Liver | 28
  Pancreas | 6
  Gastrointestinal tract | 0
  Lymph nodes | 12
  Other | 11

16. Secondary Outcome: Region-level False Negative
Description: FN regions were the regions which did not show any lesions based on [68Ga]Ga-DOTA-TATE PET/CT imaging but show at least one lesion based on CIM by central read.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Participants
  Liver | 8
  Pancreas | 8
  Gastrointestinal tract | 1
  Lymph nodes | 4
  Other | 2

17. Secondary Outcome: Region-level False Positive
Description: FP regions were the regions which showed at least one lesion based on [68Ga]Ga-DOTA-TATE PET/CT imaging but do not showed any lesion based on CIM by central read.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Participants
  Liver | 1
  Pancreas | 6
  Gastrointestinal tract | 3
  Lymph nodes | 9
  Other | 3

18. Secondary Outcome: Region-level True Negative
Description: TN regions were the regions which did not show any lesion based on both [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM by central read.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Participants
  Liver | 34
  Pancreas | 51
  Gastrointestinal tract | 67
  Lymph nodes | 46
  Other | 55

19. Secondary Outcome: Number of Participants Who Underwent a Change in Intended Treatment Plan Attributed to the [68Ga]Ga-DOTA-TATE PET/CT Imaging as Assessed by Pre and Post Imaging Questionnaires
Description: Numbers of participants for each intended treatment plan collected from physician at pre and post [68Ga]Ga-DOTA-TATE PET/CT imaging will be summarized.
Time Frame: Before and after imaging on Day 1
Population: The Efficacy Analysis Set (EFF) comprised all enrolled participants who were administered with [68Ga]Ga-DOTA-TATE. Patients with confirmed/suspected NENs had to have both results of [68Ga]Ga-DOTA-TATE PET/CT imaging and CIM, with a valid measurement without a protocol deviation with impact. Patients with confirmed/suspected NENs)
Measure: Count of Participants; unit: Participants
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 48 | 0
Participants
  Planned treatment of Chemotherapy - Before imaging | 8 |
  Planned treatment of Lutathera - Before imaging | 14 |
  Planned treatment of Observation/surveillance - Before imaging | 6 |
  Planned treatment of Radiation - Before imaging | 0 |
  Planned treatment of Somatostatin Analog - Before imaging | 15 |
  Planned treatment of Surgery - Before imaging | 5 |
  Planned treatment of Other - Before imaging | 2 |
  Planned treatment of Chemotherapy - After imaging | 6 |
  Planned treatment of Lutathera - After imaging | 17 |
  Planned treatment of Observation/surveillance - After imaging | 7 |
  Planned treatment of Radiation - After imaging | 2 |
  Planned treatment of Somatostatin Analog - After imaging | 15 |
  Planned treatment of Surgery - After imaging | 4 |
  Planned treatment of Other - After imaging | 2 |
  Participants with no change in treatment plans - After imaging | 30 |
  - Chemotherapy - After imaging | 4 |
  - Chemotherapy, Somatostatin Analog - After imaging | 2 |
  - Lutathera -After imaging | 10 |
  -Observation/surveillance -After imaging | 3 |
  - Somatostatin Analog -After imaging | 8 |
  - Surgery -After imaging | 2 |
  - Other -After imaging | 1 |
  Participants with change in treatment plans | 18 |
  -Chemotherapy Before - Lutathera After | 2 |
  -Lutathera Before - Lutathera, Radiation After | 1 |
  - Lutathera Before - Lutathera, Surgery After | 1 |
  -Lutathera Before - Observation/surveillance After | 1 |
  - Lutathera Before - Radiation After | 1 |
  - Observation/surveillance Before - Lutathera After | 1 |
  - Observation/surveillance Before - Observation/surveillance After | 1 |
  - Observation/surveillance Before - Somatostatin Analog After | 1 |
  - Somatostatin Analog Before - Lutathera After | 1 |
  - Somatostatin Analog Before - Observation/surveillance After | 1 |
  - Somatostatin Analog Before - Somatostatin Analog After | 3 |
  - Surgery Before - Lutathera, Surgery After | 1 |
  -Surgery Before - Observation/surveillance After | 1 |
  - Surgery Before - Somatostatin Analog After | 1 |
  - Other Before - Other After | 1 |

20. Secondary Outcome: Inter-reader Agreement on [68Ga]Ga-DOTA-TATE PET/CT Imaging
Description: The assessment of [68Ga]Ga-DOTA-TATE PET/CT images set was compared among the 3 independent readers.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 71
Participants
  Central Reader 1 Positive | 54
  Central Reader 2 Positive | 42
  Central Reader 3 Positive | 41
  Central Reader 1 Negative | 17
  Central Reader 2 Negative | 29
  Central Reader 3 Negative | 30

21. Secondary Outcome: Inter-reader Variability (%) on [68Ga]Ga-DOTA-TATE PET/CT Imaging
Description: Inter-reader variability for [68Ga]Ga-DOTA-TATE PET/CT imaging is defined as agreement rate among reader determinations.
  As assessed by Fleiss' Kappa statistics. Inter-reader variability (%) and its normality 95% CI is presented.
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Inter-reader variability (%)
Arm/Group | All Participants
Number analyzed (Participants) | 71
Inter-reader variability (%) | 65.2 [51.79 to 78.65]

22. Secondary Outcome: Incidence of Treatment Emergent Adverse Event (TEAE) Within 8 Days After [68Ga]Ga-DOTATATE Administration
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any occurrence of unfavorable and unintended sign(s), symptom(s) or medical condition, including abnormal laboratory findings, or worsening of any pre-existing sign(s), symptom(s) or medical condition) in a participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of any treatment used in this study. This includes events reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).
Time Frame: For treated pts: AEs are reported from the single dose of study treatment plus 8 days post treatment, up to a maximum timeframe of 9 days. For HV pts: AEs are reported from the study start plus 8 days, up to a maximum timeframe of 9 days.
Population: The Safety Set comprised all participants who received any dose of [68Ga]Ga-DOTA-TATE.
Measure: Count of Participants; unit: Participants
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 48 | 23
Participants
  Adverse events (AEs) | 8 | 2
  Adverse events - Treatment-related | 1 | 0
  Serious Adverse events (SAEs) | 2 | 0
  Serious Adverse events Treatment-related | 0 | 0
  Fatal SAEs | 0 | 0
  Fatal SAEs - Treatment-related | 0 | 0
  AEs requiring additional therapy | 3 | 0

23. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUCinf) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-inf) will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: PAS - pharmacokinetics analysis set - for treated participants with a valid measurement without a protocol deviation with impact. PK analysis was planned to be performed on a small subset of patients only, 6, and not healthy volunteers.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
h*ng/mL | 0.420 (25.5) |

24. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
h*ng/mL | 0.304 (26.3) |

25. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
ng/mL | 0.656 (30.7) |

26. Secondary Outcome: Time of Maximum Observed Drug Concentration Occurrence (Tmax) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: as for outcome 23
Measure: Median (Full Range); unit: hour
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
hour | 0.0750 [0.0333 to 0.100] |

27. Secondary Outcome: Terminal Elimination Half-life (T1/2) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
hour | 1.77 (26.3) |

28. Secondary Outcome: Total Systemic Clearance for Intravenous Administration (CL) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
L/h | 26.0 (32.5) |

29. Secondary Outcome: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz) of [68Ga]Ga-DOTA-TATE [Mass-based Concentration]
Description: Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.
Time Frame: Day 1 (5 min, 15 min, 30 min, 45 min, 60 min, 120 min, 180 min)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 6 | 0
L | 66.2 (53.5) |

30. Secondary Outcome: Lesion-level Concordance Rate for SSTR Between [68Ga]Ga-DOTA-TATE PET/CT Imaging Local Read and Local Histopathology Result Among Lesions That Local Histopathology Result Are Available
Description: The lesion-level concordance rate for SSTR between [68Ga]Ga-DOTA-TATE PET/CT imaging local read and local histopathology result among legions which is available, will be calculated. The rate is defined as the proportion of lesions which are positive or negative on both local read of [68Ga]Ga-DOTA-TATE PET/CT imaging and local histopathology among lesions detected by local histopathology.
Time Frame: Day 1 to Day 30
Population: as for outcome 9
Measure: Number; unit: lesions
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 48 | 0
lesions
  Total number of lesions with histopathology assessments | 11 |
  Positive Result of SSTR by histopathology | 8 |
  Negative Result of SSTR by histopathology | 3 |
  Positive Result of [68Ga]Ga-DOTA-TATE PET/CT imaging by local read | 11 |
  Negative Result of [68Ga]Ga-DOTA-TATE PET/CT imaging by local read | 0 |
  + Result of SSTR by histopathology - + Result of [68Ga]Ga-DOTA-TATE PET/CT imaging by local read | 8 |
  + Result of SSTR by histopathology & -Result of [68Ga]Ga-DOTA-TATE PET/CT imaging by local read | 0 |
  - Result of SSTR by histopathology & + Result of [68Ga]Ga-DOTA-TATE PET/CT imaging by local read | 3 |
  - Result of SSTR by histopathology & - Result of [68Ga]Ga-DOTA-TATE PET/CT imaging by local read | 0 |
  Lesions with concordant results | 8 |

31. Secondary Outcome: Lesion-level Concordance Rate for SSTR Between [68Ga]Ga-DOTA-TATE PET/CT Imaging Local Read and Local Histopathology Result Among Lesions That Local Histopathology Result Are Available - Concordance Rate
Description: as for outcome 30
Time Frame: Day 1 to Day 30
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Concordance rate (%)
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
Number analyzed (Participants) | 48 | 0
Concordance rate (%) | 72.7 [39.03 to 93.98] |

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the single dose of study treatment plus 8 days post treatment, up to a maximum timeframe of 9 days.
Arm/Group | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/48 | 0/23
Other Adverse Events (participants affected / at risk) | 8/48 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs (N=48) | Healthy Volunteers (N=23)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [68Ga]Ga-DOTA-TATE / Confirmed/Suspected NENs (N=48) | Healthy Volunteers (N=23)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Electrocardiogram PR prolongation (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT06240741/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT06240741/SAP_001.pdf